CLINICAL TRIAL: NCT02298205
Title: Asthma Symptom Based Adjustment of Inhaled Steroid Therapy in African American Children
Acronym: ASIST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRPO201410095
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Provider-based adjustment (Other): Primary care provider will adjust the dose of asthma controller medication based on asthma control at each encounter
  Interventions: Other: Provider-based adjustment
- Symptom-based adjustment (Active Comparator): The dose of asthma controller medication is adjusted based on the symptoms
  Interventions: Other: Asthma controller medication (Beclomethasone) adjustment strategy

INTERVENTIONS:
Other: Asthma controller medication (Beclomethasone) adjustment strategy — The participant will adjust the dose of Beclomethasone based on symptoms
  Arms: Symptom-based adjustment
Other: Provider-based adjustment — The provider will adjust the dose of Beclomethasone based on the participant's asthma control at their encounter with them
  Arms: Provider-based adjustment

SUMMARY:
African American (AA) children carry a disproportionate burden of mortality and morbidity in asthma. A major contributor to racial disparity in asthma is lack of adherence to guideline-recommended use of daily inhaled corticosteroids (ICS). Symptom-based adjustment (SBA) of ICS is a recently described patient-centered approach to asthma therapy in which patients adjust their ICS on a day-to-day basis guided by their symptoms. The overall goal of our study is to identify an acceptable, pragmatic and effective approach to asthma management in high-risk AA children. Our primary hypotheses are that SBA of ICS use is more acceptable than provider-based adjustment (PBA), equally effective in improving pediatric asthma outcomes, and will reduce the cumulative dose of ICS needed for asthma control. Therefore, in the Asthma Symptom based adjustment of Inhaled Steroid Therapy in African American children (ASIST) study, we propose a randomized, open-label, 2-arm, parallel, pragmatic trial in which we will randomly assign 200 AA children to either receive SBA or PBA for 12 months. The primary outcome is asthma control as measured by the Asthma Control Test (ACT). We propose that asthma control in the SBA group will be equivalent to the PBA group after 12 months. Secondary outcomes include monthly cumulative ICS dose, exacerbation rate, quality of life, lung function, adherence and satisfaction with the treatment plan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 6-17 years old with physician diagnosed asthma for at least 6 months
2. Self or parent reported AA Race, or mixed race with at least one grandparent with AA race
3. Receiving asthma care by the participating primary care pediatrician
4. Prescribed low dose ICS monotherapy (up to Beclomethasone 160mcg for 6-11 y/o, 240 mcg per day for over 12 year old or equivalent), or leukotriene receptor antagonist (LTRA), or low dose ICS plus LABA (for over 12 year old) for at least the past 12 weeks, regardless of adherence (see ASIST low dose ICS inclusion table for conversion of dose)
5. Asthma Evaluation Questionnaire Score (AEQ)17 0 or 1 on all 3 questions
6. Pre-BD FEV1 ≥80% of predicted
7. No history or current history of smoking
8. Ability to provide baseline information at phone screening and randomization visit
9. Ability and willingness to provide informed consent

Exclusion Criteria:

1. Pre-BD FEV1<80% of predicted within 3 months
2. Asthma requiring daily combination therapy with medium to high dose ICS with LABA
3. History of Intubation, noninvasive ventilation or ICU admission for asthma exacerbation
4. Chronic oral corticosteroid therapy
5. Chronic disease that in the opinion of the investigator/primary care provider would prevent participation in the trial
6. No landline telephone or cell phone to communicate with study staff
7. Non-English speaker
8. Another participant of ASIST in the same household

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 206 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
asthma control (change in score of asthma control test) | 12 months
  Change in score of asthma control test at 12 month from baseline

SECONDARY OUTCOMES:
Monthly cumulative dose of beclomethasone used | 12 months
Lung function (FEV1) | 12 months
  Change in lung function at 12 months compared to baseline
Patient/parent satisfaction | 12 months
  Score of satisfaction questionnaire at the end of the study
Quality of life measurement | 12 months
  Change in score in Child health survey (asthma) and PROMIS asthma questionnaire
Asthma exacerbation | 12 month
  Rate of asthma exacerbation
Missed School days | 12 months
  Number of missed school days

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States